CLINICAL TRIAL: NCT06520800
Title: Treatment and Handling Severe Obesity-Related Comorbidities in Adolescents Through Exercise
Acronym: THOR-X
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Collaborators: Lusofona University (Other)
Responsible Party: Principal Investigator, A. Videira-Silva, Professor, University of Lisbon
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THOR-X
Record Dates: First submitted 2024-07-22; First posted 2024-07-25 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Adolescent Obesity; Hypertension,Essential; Non-Alcoholic Fatty Liver Disease; Dyslipidemias; Metabolic Disease; Metabolic Syndrome
Keywords: Adolescent Obesity; Obesity treatment; Physical activity; Exercise
MeSH Terms: conditions — Pediatric Obesity; Essential Hypertension; Non-alcoholic Fatty Liver Disease; Dyslipidemias; Metabolic Diseases; Metabolic Syndrome; Motor Activity | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Series of n-of-1 trials
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Traumatic and overuse exercise-related injuries (Experimental): There is no registry of any clinically relevant adverse or unintended event associated with this kind of intervention. Nevertheless, adolescents with severe obesity may be at higher risk of both traumatic and overuse exercise-related injuries. A specific insurance for special risk participants, covering exercise-related injuries and dead (Appendix 1), will be activated in case of any adverse or unintended event during or as consequence of the exercise sessions. The impact of that specific event will be additionally analyzed and reported by the health professionals.
  Interventions: Behavioral: Treatment and handling obesity-related comorbidities in adolescents through exercise

INTERVENTIONS:
Behavioral: Treatment and handling obesity-related comorbidities in adolescents through exercise — Tailor-made, one-to-one, physical exercise program

SUMMARY:
The main objective of this project is to analyze the effect of a tailor-made, one-to-one, exercise program (aiming to treat and handle obesity-related comorbidities in adolescents with severe obesity at high risk of cardiovascular disease development) on BMI z-score, specific comorbidities, and other health-related indicators.

This project will further allow to analyze the long-term impact of the exercise program not only on clinical parameters, but also on the interaction with drug-treatment, health-related behaviors, and quality of life, further contributing to the understanding of the individual characteristics associated with a positive exercise response and frequency.

The secondary objective of the THOR-X project is to build an educational toolkit, based on project results and relevant literature, addressed to health and exercise professionals, in order to improve management of adolescents with obesity, in particular those with severe obesity.

DETAILED DESCRIPTION:
The THOR-X project is designed as a series of n-of-1 trials, with a crossover methodology. Each trial will include 3 phases and 5 assessment times organized as follows:

Phase 1. Retrospective phase. Participants/patients followed at the Pediatric Obesity Clinic (HSM, CHULN) for at least 6 months and living in Lisbon area, will be eligible for recruitment. After inclusion/exclusion criteria checking, and informed consent/assent signature, retrospective data from those who consent to participate will then be collected from clinical records. Data will be collected from the first visit and last assessments before the beginning of the intervention (baseline assessment), which will represent the control phase. The clinical records of the participants will be searched for: (i) date of first appointment, number of appointments attended, length of clinical follow-up, and emergency healthcare seeking; (ii) anthropometric and body composition data (i.e., height, weight, BMI z-score/BMI, waist and hip circumference, body fat mass, and skeletal muscle mass); (iii) clinical data (i.e., biochemical profile, blood pressure, and presence of clinical conditions, including psychopathology); (iv) physical activity and sedentary behaviors; and (v) dietary habits.

At baseline, additionally to the clinical standard assessments, the participant(s) will accomplish a battery of assessments including socio-economic, cardiorespiratory fitness, objectively measured physical activity, psycho-behavioral characteristics, sleep quality, and health-related quality of life. These assessments will allow to analyze clinical changes before intervention (control phase) and collect relevant data (not assessed previously) to better analyze intervention effect.

Phase 2. Intervention phase. The exercise intervention phase will have a 6-month duration, where participant will be exposed to two distinct exercise plans (3 months each). Per each participant, the two exercise plans will differ in terms of frequency (2 or 3 times/week), time (45 or 60 min/session) or protocol (aerobic or combined training), in a random order. Each participant will be exposed only to one exercise routine change (i.e., frequency, time, or protocol). The exercise sessions will take place at the Faculdade de Educação Física e Desporto, Universidade Lusófona. During the intervention period, the participant(s) will repeat twice (at the end of the first, and second exercise plans - 3 and 6-month) the assessments previously performed. These assessments will allow to explore the influence of exercise plan changes on the variables under study.

Phase 3. Follow-up/standard care. During the follow-up phase, the exercise-based intervention will cease, and the participant(s) will be exposed only to standard care (matching the level of exposure of phase 1 - control phase). Standard care comprises appointments with the multidisciplinary team (pediatrician, nutritionist, and exercise physiologist) every 3 months at the clinic. All the assessments performed at baseline will be repeated twice during the follow-up (12 and 18-month), which will allow to analyze short- and long-term changes associated with lack of exposure to the exercise intervention (phase 2).

ELIGIBILITY:
Inclusion Criteria:

* adolescents aged 13 to 18 years;
* of any gender (including transgender adolescents);
* with severe obesity (≥3.0 BMI z-score) [24];
* with any obesity-related comorbidity (e.g., hypertension, IR or DMT2, dyslipidemia, eating disorders, depression/anxiety);
* at least 6 months of follow-up at the Pediatric Obesity Clinic (HSM, CHULN) at the time of recruitment;
* living in Lisbon area;
* informed consent/assent signature.

Exclusion Criteria:

* major or unstable clinical conditions (other than obesity or its related comorbidities);
* inability to perform regular PA;
* pregnancy;
* mental disorders;
* smoking habits;
* being involved in another weight loss program.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI) z-score | 6 (end of intervention) and 12 months (end of follow-up)
  Calculated according to World Health Organization (WHO) data, using the WHO AnthroPlus calculator (version 1.0.4)

IPD SHARING:
Plan to Share IPD: Undecided